CLINICAL TRIAL: NCT03418649
Title: Epidural Steroid Injection With Supplemental Oral Eplerenone for Low Back Pain: A Prospective, Double Blind Randomized Trial
Brief Title: Eplerenone as a Supplement to Epidural Steroid Injections
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to recruit subjects
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Shuchita Garg, Assistant Professor of Anesthesiology & Pain Management, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017-2713
Record Dates: First submitted 2017-12-06; First posted 2018-02-01 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Degenerative Intervertebral Discs; Sciatic Radiculopathy; Low Back Pain
Keywords: low back pain; radicular pain; degenerative disc disease
MeSH Terms: conditions — Intervertebral Disc Degeneration; Low Back Pain | interventions — Eplerenone

STUDY DESIGN:
Intervention Model Description: Double blind placebo controlled. Equal numbers of subjects receive 10 day course of eplerenone or placebo following their clinically indicated epidural steroid injection
Who Masked: Participant, Care Provider, Investigator
Masking Description: Drug or look-alike placebo dispensed according to a randomization schedule.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): Eplerenone 50 Mg Tab
  Interventions: Drug: Eplerenone 50 Mg Tab
- Control (Placebo Comparator): Placebo Oral Tablet
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Eplerenone 50 Mg Tab — 50 mg PO per day for 10 days
  Other Names: Inspra
  Arms: Experimental
Drug: Placebo Oral Tablet — PO once daily for 10 days
  Other Names: placebo for eplerenone
  Arms: Control

SUMMARY:
Low back pain is a leading cause of disability and health care costs in the United States, and treatments are ineffective for many patients. Epidural steroid injections are a common treatment, but their efficacy has been questioned and for many patients they do not provide complete relief. The investigators hypothesize, based on preclinical studies, that lack of complete efficacy may be due to the fact that clinically used steroids activate not only the intended drug target, the glucocorticoid receptor, but also the pro-inflammatory mineralocorticoid receptor. To test this hypothesis, this pilot study will recruit patients scheduled for lumbar epidural steroid injections for degenerative disc disease, and randomize them to receive a concurrent treatment with oral eplerenone (a clinically approved antagonist of the mineralocorticoid receptor) or placebo for 10 days starting just after the epidural injection. At several time points during the following year, subjects will answer the Oswestry Low Back Pain Questionnaire, to report on both pain and functional outcomes.

DETAILED DESCRIPTION:
Patients with degenerative disc disease, who are recommended to have an epidural steroid injection at the participating clinics, as part of their routine clinical care, will be invited to participate in the study prior to their first epidural steroid injection. If they consent, they will complete the Oswestry Low Back Pain Questionnaire (version 2) just prior to their first injection which captures the functional effects of back pain on various activities, providing a more meaningful picture than a simple static pain rating.

The subjects will complete the Oswestry Low Back Pain Questionnaire again four weeks after their first injection, a time point at which patients routinely have a follow-up visit. Patients referred for a second injection at this time will complete an additional Oswestry just prior to that injection. Subjects will be asked to complete additional Oswestry Low Back Pain Questionnaires at 3 months, 6 months, 1 year after their epidural injection (or after their second epidural injection if this is recommended).

Prior to receiving study medication (eplerenone or placebo), subjects will provide a blood sample to examine their creatinine and potassium levels, to ensure there are no contraindications to taking eplerenone. C reactive protein levels will also be measured just prior to epidural steroid injections to determine whether this can help predict the response.

In addition to the pain questionnaires, data will be collected from the subjects' medical charts regarding basic clinical demographics and clinical outcome of the epidural steroid injection.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of lumbar degenerative disc disease demonstrated on either lumbar X-Ray or lumbar MRI.
* radicular symptoms or electromyograph consistent with radiculopathy and exam findings corresponding to this diagnosis
* Scheduled for lumbar epidural steroid injection at participating clinics as part of routine clinical care
* Negative pregnancy test, if of childbearing potential

Exclusion Criteria:

* Unable to complete questionnaires or give informed consent in English
* Unavailable for follow-up contacts to complete questionnaires
* Renal impairment (estimated glomerular filtration rate <50 mL/min or serum creatinine >1.8mg/dL) on metabolic panel obtained just prior to epidural injections.
* Elevated serum potassium (>5.5 milliequivalents/L) on metabolic panel obtained just prior to epidural injections.
* Have undergone previous lumbar surgery within the past year.
* Treated with lumbar epidural steroid injection within the past 3 months at the time of consent.
* Diabetic
* Systolic blood pressure reading less than 100 mm Hg at most recent pain clinic visit.
* Prescribed protease inhibitors.
* Taking strong CYP3A4 inhibitors
* Taking potassium supplements or potassium-sparing diuretics (amiloride, spironolactone, or triamterene) or using salt substitutes that contain potassium (examples given below and in the prescreening document to be used by the study nurse).
* Lactating.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-06 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
change in Oswestry Low Back Pain Disability Questionnaire at 12 months | Difference between score prior to and 12 months after epidural steroid injection
  back pain disability score ranging from 0 (no disability or pain) to 100% (maximum pain and disability); based on sum of responses to 10 questions each with responses ranging from 0 (no pain/disability) to 5 (maximum pain/disability) expressed as percentage of maximum score.

SECONDARY OUTCOMES:
epidural steroid injection clinical outcome | evaluated one month after injection as part of standard clinical care
  scored as 1 adequate pain relief, no further treatment recommended; 2, partial relief, second injection recommended; 3 little pain relief, alternative treatment recommended
change in Oswestry Low Back Pain Disability Questionnaire at 4 weeks | Difference between score prior to and 4 weeks after epidural steroid injection
  back pain disability score ranging from 0 (no disability or pain) to 100% (maximum pain and disability); based on sum of responses to 10 questions each with responses ranging from 0 (no pain/disability) to 5 (maximum pain/disability) expressed as percentage of maximum score.
change in Oswestry Low Back Pain Disability Questionnaire at 3 months | Difference between score prior to and 3 months after epidural steroid injection
  back pain disability score ranging from 0 (no disability or pain) to 100% (maximum pain and disability); based on sum of responses to 10 questions each with responses ranging from 0 (no pain/disability) to 5 (maximum pain/disability) expressed as percentage of maximum score.
change in Oswestry Low Back Pain Disability Questionnaire at 6 months | Difference between score prior to and 6 months after epidural steroid injection
  back pain disability score ranging from 0 (no disability or pain) to 100% (maximum pain and disability); based on sum of responses to 10 questions each with responses ranging from 0 (no pain/disability) to 5 (maximum pain/disability) expressed as percentage of maximum score.

CONTACTS AND LOCATIONS:
Overall Officials: Shuchita Garg, MD, Principal Investigator — University of Cincinnati
Locations (2):
- United States (2):
  - UC Health Pain Medicine Center in Clifton, Cincinnati, Ohio
  - UC Health Pain Medicine Center in West Chester, West Chester, Ohio

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2017-08-22): https://cdn.clinicaltrials.gov/large-docs/49/NCT03418649/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-17): https://cdn.clinicaltrials.gov/large-docs/49/NCT03418649/SAP_001.pdf